CLINICAL TRIAL: NCT04784832
Title: Transcranial Magnetic Stimulation-based Assessment of Mental Training Effects on Motor Learning in Healthy Participants
Brief Title: TMS-based Assessment of Mental Training Effects on Motor Learning in Healthy Participants
Acronym: IMAP-TMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: C19-19; 2020-A00305-34 / 1 (Registry Identifier: IDRCB)
Record Dates: First submitted 2020-12-07; First posted 2021-03-05 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Motor Learning
MeSH Terms: interventions — Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation; Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (28):
- Sequence 1 - Training with same task - Long follow-up (Experimental): Motor task (Pretest and Posttests on the same task) Transcranial magnetic stimulation Mental training
  Interventions: Device: Transcranial magnetic stimulation; Other: Mental training
- Sequence 1 - Training with same task - Short follow-up (Experimental): Motor task (Pretest and Posttests on the same task) Transcranial magnetic stimulation Mental training
  Interventions: Device: Transcranial magnetic stimulation; Other: Mental training
- Sequence 1 - Training with different tasks - Long follow-up (Experimental): Motor task (different task in immediate post test) Transcranial magnetic stimulation Mental training
  Interventions: Device: Transcranial magnetic stimulation; Other: Mental training
- Sequence 1 - Training with different tasks - Short follow-up (Experimental): Motor task (different task in immediate post test) Transcranial magnetic stimulation Mental training
  Interventions: Device: Transcranial magnetic stimulation; Other: Mental training
- Sequence 1 - Training with muscle contractions - Long follow-up (Experimental): Motor task (isometric muscle contractions in immediate post test) Transcranial magnetic stimulation Mental training
  Interventions: Device: Transcranial magnetic stimulation; Other: Mental training
- Sequence 1 - Training with muscle contractions - Short follow-up (Experimental): Motor task (isometric muscle contractions in immediate post test) Transcranial magnetic stimulation Mental training
  Interventions: Device: Transcranial magnetic stimulation; Other: Mental training
- Sequence 1 - Control (Active Comparator): Motor task (Pretest and Posttests on the same task) Transcranial magnetic stimulation No mental training
  Interventions: Device: Transcranial magnetic stimulation
- Sequence 2 - Physical training with perturbation during preparation - Long follow-up (Active Comparator): Motor task (Pretest and Posttests) Transcranial magnetic stimulation External pertubation (robotic arm) Physical training
  Interventions: Device: Transcranial magnetic stimulation; Device: Robotic arm; Other: Physical training
- Sequence 2 - Physical training with perturbation during preparation - Short follow-up (Active Comparator): Motor task (Pretest and Posttests) Transcranial magnetic stimulation External pertubation (robotic arm) Physical training
  Interventions: Device: Transcranial magnetic stimulation; Device: Robotic arm; Other: Physical training
- Sequence 2 - Physical training with perturbation after preparation - Long follow-up (Active Comparator): Motor task (Pretest and Posttests) Transcranial magnetic stimulation External pertubation (robotic arm) Physical training
  Interventions: Device: Transcranial magnetic stimulation; Device: Robotic arm; Other: Physical training
- Sequence 2 - Physical training with perturbation after preparation - Short follow-up (Active Comparator): Motor task (Pretest and Posttests) Transcranial magnetic stimulation External pertubation (robotic arm) Physical training
  Interventions: Device: Transcranial magnetic stimulation; Device: Robotic arm; Other: Physical training
- Sequence 2 - Mental training with perturbation during preparation - Long follow-up (Experimental): Motor task (Pretest and Posttests) Transcranial magnetic stimulation External pertubation (robotic arm) Mental training
  Interventions: Device: Transcranial magnetic stimulation; Device: Robotic arm; Other: Mental training
- Sequence 2 - Mental training with perturbation during preparation - Short follow-up (Experimental): Motor task (Pretest and Posttests) Transcranial magnetic stimulation External pertubation (robotic arm) Mental training
  Interventions: Device: Transcranial magnetic stimulation; Device: Robotic arm; Other: Mental training
- Sequence 2 - Mental training with perturbation after preparation - Long follow-up (Experimental): Motor task (Pretest and Posttests) Transcranial magnetic stimulation External pertubation (robotic arm) Mental training
  Interventions: Device: Transcranial magnetic stimulation; Device: Robotic arm; Other: Mental training
- Sequence 2 - Mental training with perturbation after preparation - Short follow-up (Experimental): Motor task (Pretest and Posttests) Transcranial magnetic stimulation External pertubation (robotic arm) Mental training
  Interventions: Device: Transcranial magnetic stimulation; Device: Robotic arm; Other: Mental training
- Sequence 3 - Training (same task) - Long follow-up (Experimental): Paired Associative Stimulation Mental training (same as the motor task) Motor task Transcranial magnetic stimulation Peripheral nerve stimulation Cervicomedullar stimulation
  Interventions: Device: Transcranial magnetic stimulation; Device: Peripheral Nerve Stimulation; Device: Paired Associative Stimulation; Device: Cervicomedullar stimulation; Other: Mental training
- Sequence 3 - Training (same task) - Short follow-up (Experimental): Paired Associative Stimulation Mental training (same as the motor task) Motor task Transcranial magnetic stimulation Peripheral nerve stimulation Cervicomedullar stimulation
  Interventions: Device: Transcranial magnetic stimulation; Device: Peripheral Nerve Stimulation; Device: Paired Associative Stimulation; Device: Cervicomedullar stimulation; Other: Mental training
- Sequence 3 - Training (different task) - Long follow-up (Experimental): Paired Associative Stimulation Mental training (different of the motor task) Motor task Transcranial magnetic stimulation Peripheral nerve stimulation Cervicomedullar stimulation
  Interventions: Device: Transcranial magnetic stimulation; Device: Peripheral Nerve Stimulation; Device: Paired Associative Stimulation; Device: Cervicomedullar stimulation; Other: Mental training
- Sequence 3 - Training (different task) - Short follow-up (Experimental): Paired Associative Stimulation Mental training (different of the motor task) Motor task Transcranial magnetic stimulation Peripheral nerve stimulation Cervicomedullar stimulation
  Interventions: Device: Transcranial magnetic stimulation; Device: Peripheral Nerve Stimulation; Device: Paired Associative Stimulation; Device: Cervicomedullar stimulation; Other: Mental training
- Sequence 3 - Control 1 (Active Comparator): Mental Training Motor task (same as the motor task) Transcranial magnetic stimulation Peripheral nerve stimulation Cervicomedullar stimulation
  Interventions: Device: Transcranial magnetic stimulation; Device: Peripheral Nerve Stimulation; Device: Cervicomedullar stimulation; Other: Mental training
- Sequence 3 - Control 2 (Active Comparator): Paired Associative Stimulation Motor task Transcranial magnetic stimulation Peripheral nerve stimulation Cervicomedullar stimulation
  Interventions: Device: Transcranial magnetic stimulation; Device: Peripheral Nerve Stimulation; Device: Paired Associative Stimulation; Device: Cervicomedullar stimulation
- Sequence 4 - Immobilization - Short follow-up (Experimental): Transcranial magnetic stimulation Arm immobilization Motor task Mental training
  Interventions: Device: Transcranial magnetic stimulation; Device: Wrist; Other: Mental training
- Sequence 4 - Immobilization - Long follow-up (Experimental): Transcranial magnetic stimulation Arm immobilization Motor task Mental training
  Interventions: Device: Transcranial magnetic stimulation; Device: Wrist; Other: Mental training
- Sequence 4 - Cathodal - Short follow-up (Experimental): Transcranial magnetic stimulation Cathodal transcranial direct current stimulation Motor task Mental training
  Interventions: Device: Transcranial magnetic stimulation; Device: Transcranial direct current stimulation; Other: Mental training
- Sequence 4 - Cathodal - Long follow-up (Experimental): Transcranial magnetic stimulation Cathodal transcranial direct current stimulation Motor task Mental training
  Interventions: Device: Transcranial magnetic stimulation; Device: Transcranial direct current stimulation; Other: Mental training
- Sequence 4 - Anodal - Short follow-up (Experimental): Transcranial magnetic stimulation Anodal transcranial direct current stimulation Motor task Mental training
  Interventions: Device: Transcranial magnetic stimulation; Device: Transcranial direct current stimulation; Other: Mental training
- Sequence 4 - Anodal - Long follow-up (Experimental): Transcranial magnetic stimulation Anodal transcranial direct current stimulation Motor task Mental training
  Interventions: Device: Transcranial magnetic stimulation; Device: Transcranial direct current stimulation; Other: Mental training
- Sequence 4 - Control (Sham Comparator): Transcranial magnetic stimulation Motor task Mental training
  Interventions: Device: Transcranial magnetic stimulation; Other: Mental training

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Magnetic stimulation of the cortex
  Other Names: TMS
Device: Peripheral Nerve Stimulation — Electric stimulation of the nerves
  Arms: Sequence 3 - Control 1; Sequence 3 - Control 2; Sequence 3 - Training (different task) - Long follow-up; Sequence 3 - Training (different task) - Short follow-up; Sequence 3 - Training (same task) - Long follow-up; Sequence 3 - Training (same task) - Short follow-up
Device: Transcranial direct current stimulation — Electric stimulation of the cortex
  Other Names: tDCS
  Arms: Sequence 4 - Anodal - Long follow-up; Sequence 4 - Anodal - Short follow-up; Sequence 4 - Cathodal - Long follow-up; Sequence 4 - Cathodal - Short follow-up
Device: Paired Associative Stimulation — Combined magnetic and electric stimulation of cortex and nerve, respectively
  Other Names: PAS
  Arms: Sequence 3 - Control 2; Sequence 3 - Training (different task) - Long follow-up; Sequence 3 - Training (different task) - Short follow-up; Sequence 3 - Training (same task) - Long follow-up; Sequence 3 - Training (same task) - Short follow-up
Device: Wrist — Short-term immobilization of the arm
  Arms: Sequence 4 - Immobilization - Long follow-up; Sequence 4 - Immobilization - Short follow-up
Device: Robotic arm — External perturbation of force field induced by robotic arm
  Arms: Sequence 2 - Mental training with perturbation after preparation - Long follow-up; Sequence 2 - Mental training with perturbation after preparation - Short follow-up; Sequence 2 - Mental training with perturbation during preparation - Long follow-up; Sequence 2 - Mental training with perturbation during preparation - Short follow-up; Sequence 2 - Physical training with perturbation after preparation - Long follow-up; Sequence 2 - Physical training with perturbation after preparation - Short follow-up; Sequence 2 - Physical training with perturbation during preparation - Long follow-up; Sequence 2 - Physical training with perturbation during preparation - Short follow-up
Device: Cervicomedullar stimulation — Electric stimulation of the muscle
  Arms: Sequence 3 - Control 1; Sequence 3 - Control 2; Sequence 3 - Training (different task) - Long follow-up; Sequence 3 - Training (different task) - Short follow-up; Sequence 3 - Training (same task) - Long follow-up; Sequence 3 - Training (same task) - Short follow-up
Other: Physical training — Training to perform the task by actually doing the task
  Arms: Sequence 2 - Physical training with perturbation after preparation - Long follow-up; Sequence 2 - Physical training with perturbation after preparation - Short follow-up; Sequence 2 - Physical training with perturbation during preparation - Long follow-up; Sequence 2 - Physical training with perturbation during preparation - Short follow-up
Other: Mental training — Training to perform the task by imaging doing the task
  Arms: Sequence 1 - Training with different tasks - Long follow-up; Sequence 1 - Training with different tasks - Short follow-up; Sequence 1 - Training with muscle contractions - Long follow-up; Sequence 1 - Training with muscle contractions - Short follow-up; Sequence 1 - Training with same task - Long follow-up; Sequence 1 - Training with same task - Short follow-up; Sequence 2 - Mental training with perturbation after preparation - Long follow-up; Sequence 2 - Mental training with perturbation after preparation - Short follow-up; Sequence 2 - Mental training with perturbation during preparation - Long follow-up; Sequence 2 - Mental training with perturbation during preparation - Short follow-up; Sequence 3 - Control 1; Sequence 3 - Training (different task) - Long follow-up; Sequence 3 - Training (different task) - Short follow-up; Sequence 3 - Training (same task) - Long follow-up; Sequence 3 - Training (same task) - Short follow-up; Sequence 4 - Anodal - Long follow-up; Sequence 4 - Anodal - Short follow-up; Sequence 4 - Cathodal - Long follow-up; Sequence 4 - Cathodal - Short follow-up; Sequence 4 - Control; Sequence 4 - Immobilization - Long follow-up; Sequence 4 - Immobilization - Short follow-up

SUMMARY:
The general purpose of this research project is to analyze the specific role of motor imagery on motor learning, assessed through corticospinal excitability measurements and behavioral data collection. This project is based on four sequences. For Sequence 1, the main objective is to examine the effect of mental training on movement speed and accuracy in a manual motor sequence task, as well as the influence of sensory feedback in immediate post-test (i.e., execution of a similar, but not identical, manual motor sequence, other manual tasks) on performance in delayed post-test. The secondary objective will be to examine corticospinal changes (i.e., amplitude of motor evoked potentials) induced by mental training, by measuring the amplitude of motor evoked potentials before and after mental training. For Sequence 2, the main objective is to examine the impact of a motor disturbance induced by a robotic arm at different intervals during the motor imagery process. The secondary objective will be to examine the corticospinal changes (i.e. amplitude of evoked motor potentials) induced by mental training as a function of the applied perturbations, before and after perturbation. For Sequence 3, the main objective will be to examine the influence of neuroplasticity on the quality of mental training. More specifically, the investigators will study the links between brain plasticity and motor learning through mental training. The secondary objective will be to examine the corticospinal changes (i.e. amplitude of evoked motor potentials) induced by mental training at different levels of the neuromuscular system (cortical, cervicomedullar, peripheral) after a training period. For Sequence 4, the main objective will be to examine the effect of short-term arm-immobilization of on the retention of motor learning induced by mental training. The secondary objective will be to examine the corticospinal changes (i.e., amplitude of motor evoked potentials) induced by of short-term arm-immobilization, or by transcranial direct current stimulation (tDCS), on motor learning. The results of this fundamental research project will allow a better understanding of neurophysiological and behavioral mechanisms that underlie motor learning through motor imagery. The results will allow to efficiently consider inter-individual specificities and will thus open up to clinical research perspectives, towards the establishment of adapted motor rehabilitation protocols.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 60 years old
* Having given written informed consent
* Affiliated to a social security scheme

Exclusion Criteria:

* History of psychiatric illness (declarative)
* Person under guardianship, curatorship, safeguard of justice
* Neurological problem that could bias the results of the study (declarative)
* Personal or family history of epilepsy
* Person deprived of liberty by judicial or administrative decision
* Person hospitalized without consent and not subject to legal protection, and person admitted to a health or social institution for purposes other than that of the research
* Person subject to an exclusion period for another research
* Pregnant women or women of childbearing age not using known contraception
* Breastfeeding women
* Person on medication that could influence neurophysiological measures (neuroleptics, anxiolytics, antidepressants)
* Person carrying :
* pacemaker or other device that could interfere with the magnetic field
* Implants (mechanical or electronic: cochlear implants, neural or cardiac pacemakers, infusion pumps, magnetic aneurysm clips, etc.)
* Metallic foreign bodies in the eye or nervous system
* Metallic objects (tattoos, piercings, etc.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 556 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2027-04-07 (Estimated); Study Completion 2027-04-07 (Estimated)

PRIMARY OUTCOMES:
Evolution of movement speed - Sequence 1 | Each day in Sequence 1 (Sequence 1 is 11 days)
  The duration of performed movement sequences
Evolution of movement accuracy - Sequence 1 | Each day in Sequence 1 (Sequence 1 is 11 days)
  The accuracy of performed movement sequences (i.e., the correspondence between the performed finger motor sequences and the requested finger motor sequence).
Evolution of trajectory error - Sequence 2 | Each day in Sequence 2 (Sequence 1 is 10 days)
  The area under the curve of hand's trajectory according to the straight line joining the starting target and the final target.
Evolution of maximal deviation - Sequence 2 | Each day in Sequence 2 (Sequence 1 is 10 days)
  The maximal perpendicular distance between the position of the hand and the straight line joining the starting target and the final target
Evolution of final error - Sequence 2 | Each day in Sequence 2 (Sequence 1 is 10 days)
  The distance between the final position of the hand and the position of the final target.
Evolution of movement speed - Sequence 3 | Each day from day 2 to day 11 of Sequence 3 (Sequence 3 is 11 days)
  The duration of performed movement sequences
Evolution of movement accuracy - Sequence 3 | Each day from day 2 to day 11 of Sequence 3 (Sequence 3 is 11 days)
  The accuracy of performed movement sequences (i.e., the correspondence between the performed finger motor sequences and the requested finger motor sequence).
Evolution of movement speed - Sequence 4 | Each day in Sequence 4 (Sequence 4 is 6 days)
  The duration of performed movement sequences
Evolution of movement accuracy - Sequence 4 | Each day in Sequence 4 (Sequence 4 is 6 days)
  The accuracy of performed movement sequences (i.e., the correspondence between the performed finger motor sequences and the requested finger motor sequence).

SECONDARY OUTCOMES:
Evolution of motor evoked potentials amplitude - Sequence 1 | Day 1, 5, 6, 10 and 11 in Sequence 1 (Sequence 1 is 11 days).
  Peak-to-peak amplitude of motor evoked potentials
Evolution of motor evoked potentials amplitude - Sequence 2 | Each day in Sequence 2 (Sequence 2 is 10 days)
  Peak-to-peak amplitude of motor evoked potentials
Evolution of motor evoked potentials amplitude - Sequence 3 | Day 1, 5, 6, 10 and 11 in Sequence 3 (Sequence 1 is 11 days)
  Peak-to-peak amplitude of motor evoked potentials
Evolution of motor evoked potentials amplitude - Sequence 4 | Days 1, 5, and 6 in Sequence 4 (Sequence 4 is 6 days)
  Peak-to-peak amplitude of motor evoked potentials

CONTACTS AND LOCATIONS:
Overall Officials: Florent Lebon, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- INSERM - U1093 Cognition, Action, and Sensorimotor Plasticity, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abraham WC. Metaplasticity: tuning synapses and networks for plasticity. Nat Rev Neurosci. 2008 May;9(5):387. doi: 10.1038/nrn2356. PMID 18401345
- [Background] Anwar MN, Khan SH. Trial-by-trial adaptation of movements during mental practice under force field. Comput Math Methods Med. 2013;2013:109497. doi: 10.1155/2013/109497. Epub 2013 May 7. PMID 23737857
- [Background] Allami N, Paulignan Y, Brovelli A, Boussaoud D. Visuo-motor learning with combination of different rates of motor imagery and physical practice. Exp Brain Res. 2008 Jan;184(1):105-13. doi: 10.1007/s00221-007-1086-x. Epub 2007 Sep 12. PMID 17849109
- [Background] Arora S, Aggarwal R, Sevdalis N, Moran A, Sirimanna P, Kneebone R, Darzi A. Development and validation of mental practice as a training strategy for laparoscopic surgery. Surg Endosc. 2010 Jan;24(1):179-87. doi: 10.1007/s00464-009-0624-y. Epub 2009 Jul 25. PMID 19633892
- [Background] Avanzino L, Giannini A, Tacchino A, Pelosin E, Ruggeri P, Bove M. Motor imagery influences the execution of repetitive finger opposition movements. Neurosci Lett. 2009 Nov 27;466(1):11-5. doi: 10.1016/j.neulet.2009.09.036. Epub 2009 Sep 20. PMID 19770024
- [Background] Bienenstock EL, Cooper LN, Munro PW. Theory for the development of neuron selectivity: orientation specificity and binocular interaction in visual cortex. J Neurosci. 1982 Jan;2(1):32-48. doi: 10.1523/JNEUROSCI.02-01-00032.1982. PMID 7054394
- [Background] Burianova H, Marstaller L, Sowman P, Tesan G, Rich AN, Williams M, Savage G, Johnson BW. Multimodal functional imaging of motor imagery using a novel paradigm. Neuroimage. 2013 May 1;71:50-8. doi: 10.1016/j.neuroimage.2013.01.001. Epub 2013 Jan 12. PMID 23319043
- [Background] Cantarero G, Tang B, O'Malley R, Salas R, Celnik P. Motor learning interference is proportional to occlusion of LTP-like plasticity. J Neurosci. 2013 Mar 13;33(11):4634-41. doi: 10.1523/JNEUROSCI.4706-12.2013. PMID 23486938
- [Background] Classen J, Liepert J, Wise SP, Hallett M, Cohen LG. Rapid plasticity of human cortical movement representation induced by practice. J Neurophysiol. 1998 Feb;79(2):1117-23. doi: 10.1152/jn.1998.79.2.1117. PMID 9463469
- [Background] Cumming J, Hall C. Deliberate imagery practice: the development of imagery skills in competitive athletes. J Sports Sci. 2002 Feb;20(2):137-45. doi: 10.1080/026404102317200846. PMID 11811570
- [Background] Decety J. The neurophysiological basis of motor imagery. Behav Brain Res. 1996 May;77(1-2):45-52. doi: 10.1016/0166-4328(95)00225-1. PMID 8762158
- [Background] Doyon J, Bellec P, Amsel R, Penhune V, Monchi O, Carrier J, Lehericy S, Benali H. Contributions of the basal ganglia and functionally related brain structures to motor learning. Behav Brain Res. 2009 Apr 12;199(1):61-75. doi: 10.1016/j.bbr.2008.11.012. Epub 2008 Nov 17. PMID 19061920
- [Background] Doyon J, Benali H. Reorganization and plasticity in the adult brain during learning of motor skills. Curr Opin Neurobiol. 2005 Apr;15(2):161-7. doi: 10.1016/j.conb.2005.03.004. PMID 15831397
- [Background] Gentili R, Han CE, Schweighofer N, Papaxanthis C. Motor learning without doing: trial-by-trial improvement in motor performance during mental training. J Neurophysiol. 2010 Aug;104(2):774-83. doi: 10.1152/jn.00257.2010. Epub 2010 Jun 10. PMID 20538766
- [Background] Gentili R, Papaxanthis C, Pozzo T. Improvement and generalization of arm motor performance through motor imagery practice. Neuroscience. 2006 Feb;137(3):761-72. doi: 10.1016/j.neuroscience.2005.10.013. Epub 2005 Dec 9. PMID 16338093
- [Background] Grush R. The emulation theory of representation: motor control, imagery, and perception. Behav Brain Sci. 2004 Jun;27(3):377-96; discussion 396-442. doi: 10.1017/s0140525x04000093. PMID 15736871
- [Background] Guillot A, Moschberger K, Collet C. Coupling movement with imagery as a new perspective for motor imagery practice. Behav Brain Funct. 2013 Feb 20;9:8. doi: 10.1186/1744-9081-9-8. PMID 23425312
- [Background] Halsband U, Lange RK. Motor learning in man: a review of functional and clinical studies. J Physiol Paris. 2006 Jun;99(4-6):414-24. doi: 10.1016/j.jphysparis.2006.03.007. Epub 2006 May 26. PMID 16730432
- [Background] Izawa J, Shadmehr R. Learning from sensory and reward prediction errors during motor adaptation. PLoS Comput Biol. 2011 Mar;7(3):e1002012. doi: 10.1371/journal.pcbi.1002012. Epub 2011 Mar 10. PMID 21423711
- [Background] Jeannerod M. Neural simulation of action: a unifying mechanism for motor cognition. Neuroimage. 2001 Jul;14(1 Pt 2):S103-9. doi: 10.1006/nimg.2001.0832. PMID 11373140
- [Background] Karni A, Meyer G, Jezzard P, Adams MM, Turner R, Ungerleider LG. Functional MRI evidence for adult motor cortex plasticity during motor skill learning. Nature. 1995 Sep 14;377(6545):155-8. doi: 10.1038/377155a0. PMID 7675082
- [Background] Keller PE. Mental imagery in music performance: underlying mechanisms and potential benefits. Ann N Y Acad Sci. 2012 Apr;1252:206-13. doi: 10.1111/j.1749-6632.2011.06439.x. PMID 22524361
- [Background] Lebon F, Lotze M, Stinear CM, Byblow WD. Task-dependent interaction between parietal and contralateral primary motor cortex during explicit versus implicit motor imagery. PLoS One. 2012;7(5):e37850. doi: 10.1371/journal.pone.0037850. Epub 2012 May 31. PMID 22693579
- [Background] Lehericy S, Benali H, Van de Moortele PF, Pelegrini-Issac M, Waechter T, Ugurbil K, Doyon J. Distinct basal ganglia territories are engaged in early and advanced motor sequence learning. Proc Natl Acad Sci U S A. 2005 Aug 30;102(35):12566-71. doi: 10.1073/pnas.0502762102. Epub 2005 Aug 17. PMID 16107540
- [Background] Malouin F, Jackson PL, Richards CL. Towards the integration of mental practice in rehabilitation programs. A critical review. Front Hum Neurosci. 2013 Sep 19;7:576. doi: 10.3389/fnhum.2013.00576. PMID 24065903
- [Background] Minkova L, Peter J, Abdulkadir A, Schumacher LV, Kaller CP, Nissen C, Kloppel S, Lahr J. Determinants of Inter-Individual Variability in Corticomotor Excitability Induced by Paired Associative Stimulation. Front Neurosci. 2019 Aug 14;13:841. doi: 10.3389/fnins.2019.00841. eCollection 2019. PMID 31474818
- [Background] Mulder T. Motor imagery and action observation: cognitive tools for rehabilitation. J Neural Transm (Vienna). 2007;114(10):1265-78. doi: 10.1007/s00702-007-0763-z. Epub 2007 Jun 20. PMID 17579805
- [Background] Opie GM, Evans A, Ridding MC, Semmler JG. Short-term immobilization influences use-dependent cortical plasticity and fine motor performance. Neuroscience. 2016 Aug 25;330:247-56. doi: 10.1016/j.neuroscience.2016.06.002. Epub 2016 Jun 6. PMID 27282084
- [Background] Palmiero M, Belardinelli MO, Nardo D, Sestieri C, Di Matteo R, D'Ausilio A, Romani GL. Mental imagery generation in different modalities activates sensory-motor areas. Cogn Process. 2009 Sep;10 Suppl 2:S268-71. doi: 10.1007/s10339-009-0324-5. No abstract available. PMID 19693586
- [Background] Rozand V, Lebon F, Stapley PJ, Papaxanthis C, Lepers R. A prolonged motor imagery session alter imagined and actual movement durations: Potential implications for neurorehabilitation. Behav Brain Res. 2016 Jan 15;297:67-75. doi: 10.1016/j.bbr.2015.09.036. Epub 2015 Sep 30. PMID 26431764
- [Background] Rosenkranz K, Seibel J, Kacar A, Rothwell J. Sensorimotor deprivation induces interdependent changes in excitability and plasticity of the human hand motor cortex. J Neurosci. 2014 May 21;34(21):7375-82. doi: 10.1523/JNEUROSCI.5139-13.2014. PMID 24849369
- [Background] Ruffino C, Papaxanthis C, Lebon F. The influence of imagery capacity in motor performance improvement. Exp Brain Res. 2017 Oct;235(10):3049-3057. doi: 10.1007/s00221-017-5039-8. Epub 2017 Jul 21. PMID 28733754
- [Background] Saimpont A, Mercier C, Malouin F, Guillot A, Collet C, Doyon J, Jackson PL. Anodal transcranial direct current stimulation enhances the effects of motor imagery training in a finger tapping task. Eur J Neurosci. 2016 Jan;43(1):113-9. doi: 10.1111/ejn.13122. Epub 2015 Dec 15. PMID 26540137
- [Background] Rulleau T, Robin N, Abou-Dest A, Chesnet D, Toussaint L. Does the Improvement of Position Sense Following Motor Imagery Practice Vary as a Function of Age and Time of Day? Exp Aging Res. 2018 Oct-Dec;44(5):443-454. doi: 10.1080/0361073X.2018.1521496. Epub 2018 Oct 9. PMID 30300100
- [Background] Schuster C, Hilfiker R, Amft O, Scheidhauer A, Andrews B, Butler J, Kischka U, Ettlin T. Best practice for motor imagery: a systematic literature review on motor imagery training elements in five different disciplines. BMC Med. 2011 Jun 17;9:75. doi: 10.1186/1741-7015-9-75. PMID 21682867

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT04784832/Prot_SAP_000.pdf